CLINICAL TRIAL: NCT05957536
Title: A Phase 1, Open-label Dose Escalation and Dose-Expansion Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of D3L-001 Monotherapy in Subjects With HER2-Positive Advanced Solid Tumors.
Brief Title: A Study of D3L-001 as Monotherapy in Subjects With HER2-Positive Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: D3 Bio (Wuxi) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D3L-001-100
Record Dates: First submitted 2023-07-07; First posted 2023-07-24 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: HER-2 Positive Advanced Solid Tumors
Keywords: HER-2 Positive; Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- D3L-001 (Experimental): Part 1 Dose Escalation in subjects with HER2-positive advanced solid tumors
  * Cohort 1 (starting dose)
  * Cohort 2
  * Cohort 3
  * Cohort 4
  * Cohort 5
  Part 2 Dose Expansion
  * Cohort A for subjects with HER2-positive advanced breast cancer
  * Cohort B for subjects with HER2-positive advanced gastric cancer/gastroesophageal junction cancer
  Interventions: Biological: D3L-001

INTERVENTIONS:
Biological: D3L-001 — Intravenous administration

SUMMARY:
This first-in-human (FIH) study, multi-center, open-label, dose escalation and dose expansion Phase I study to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), immunogenicity, and preliminary anti-tumor activity of D3L-001 in subjects with HER2-positive advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have documented HER2 positivity (determined by immunohistochemistry [IHC], in situ hybridization [ISH], Next Generation Sequencing [NGS] or other analysis techniques as appropriate).
* Subject must have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Subject must have left ventricular ejection fraction (LVEF) ≥50% by either echocardiography (ECHO) or multiple-gated acquisition (MUGA) within the screening period.
* Subject must have adequate organ and marrow function within the screening period.

Exclusion Criteria:

* Subject has any prior treatment with anti-CD47 or SIRPα agent.
* Subject has major surgery or radiotherapy, immunostimulatory agents, investigational agents, or any other anticancer treatment including chemotherapy, targeted therapy, biologics that is not completed 28 days before first dose of study medication.
* Subject has immunosuppressive medication that is not completed 14 days before the first dose of study medication.
* Subject has uncontrolled intercurrent illness that would limit compliance with study requirements, substantially increase risk of incurring AEs, or compromise the ability of the subject to give written informed consent.
* Subject has unresolved treatment-related toxicities from previous anticancer therapy of NCI CTCAE Grade ≥2 (with exception of vitiligo or alopecia).
* Judgment by the Investigator that the subject should not participate in the study if the subject is unlikely to comply with study procedures, restrictions, and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2026-03-11 (Estimated); Study Completion 2026-03-11 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Screening until Safety Follow Up visit (30 days after the last dose)
Maximum Tolerated Dose based on Dose-Limiting Toxicities (DLTs) | At the end of Cycle 1 (each cycle is 21 days).

SECONDARY OUTCOMES:
D3L-001 minimum serum concentration (Ctrough) | First dose up to 6 months
D3L-001 maximum observed plasma concentration (Cmax) | First dose up to 6 months
D3L-001 time to maximum plasma concentration (tmax) | First dose up to 6 months
D3L-001 half-life (t1/2) | First dose up to 6 months
D3L-001 area under the concentration-time curve (AUC) | First dose up to 6 months
Incidence of anti-drug antibodies (ADA) to D3L-001 | First dose up to 6 months
Objective response rate (ORR) as Determined by the Investigator According to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1) | Until disease progression or end of treatment (up to approximately 24 months)
Duration of Response (DOR) as Determined by the Investigator According to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1) | Until disease progression or end of treatment (up to approximately 24 months)
Disease control rate (DCR) as Determined by the Investigator According to Response Evaluation Criteria in Solid Tumors, Version 1.1 | Until disease progression or end of treatment (up to approximately 24 months)
Progression-free survival (PFS) as determined by the investigator according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1) | Until disease progression or end of treatment (up to approximately 24 months)
Pre- and post-dose levels of CD47 receptor occupancy in particular cell types from peripheral blood | First dose up to 6 months

CONTACTS AND LOCATIONS:
Locations (9):
- United States (4):
  - D3 Bio Investigative Site, Stanford, California
  - D3 Bio Investigative Site, Boston, Massachusetts
  - D3 Bio Investigative Site, New York, New York
  - D3 Bio Investigative Site, San Antonio, Texas
- Australia (2):
  - D3 Bio Investigative Site, Sydney, New South Wales
  - D3 Bio Investigative Site, Malvern, Victoria
- China (3):
  - D3 Bio Investigative Site, Harbin, Heilongjiang
  - D3 Bio Investigative Site, Shanghai, Shanghai Municipality
  - D3 Bio Investigative Site, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No